CLINICAL TRIAL: NCT01906450
Title: STUDY ON THE EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER HIGH SENSITIVE C-REACTIVE PROTEIN. RANDOMIZED CONTROLLED CLINICAL TRIAL.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Responsible Party: Principal Investigator, Jorge Enrique Soto, periodontist Cert. DDS, Universidad del Valle, Colombia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL1688
Record Dates: First submitted 2013-05-23; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Scaling and root planing plus Azithromycin (Experimental): Single session of scaling and root planning. Azithromycin tablets 500mg, 1 tablet every 24 hours for 5 days
  Interventions: Drug: Scaling and root planing plus Azithromycin
- Scaling and root planing plus placebo (Placebo Comparator): Single session of scaling and root planning placebo tablets 500mg, 1 tablet every 24 hours for 3 days
  Interventions: Drug: Scaling and root planing plus placebo
- baselline screening only (No Intervention): Dental prophylaxis is offered

INTERVENTIONS:
Drug: Scaling and root planing plus Azithromycin — Single session of scaling and root planning using ultrasonic device. Azithromycin tablets 500mg, 1 tablet every 24 hours for 5 days
  Arms: Scaling and root planing plus Azithromycin
Drug: Scaling and root planing plus placebo — Single session of scaling and root planning placebo tablets 500mg, 1 tablet every 24 hours for 3 days
  Arms: Scaling and root planing plus placebo

SUMMARY:
Human periodontitis is a group of highly prevalent oral inflammatory diseases and infections with relatively easy treatment and preventive features. The present study is aimed to determine if treating human individuals with chronic periodontitis, along with the use of antibiotics, reduces cardiovascular risk marker (HsPCR) and also intends to identify if severity of periodontitis could be associated with a raise of systemic inflammatory biomarkers on baseline.

ELIGIBILITY:
Inclusion Criteria:

* must be of legal age (≥ 18 years old)
* voluntary participation and signed information consent
* confirmed systemically healthy individual
* at least 15 teeth present in mouth

Exclusion Criteria

* pregnant women
* smokers
* antibiotic consumption 6 months before inclusion
* HIV positive or AIDS
* Allergic reactions to macrolides and specifically to azithromycin
* Periodontal treatment 6 months before inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER HIGH SENSITIVE C-REACTIVE PROTEIN. | 3 months
  High sensitive C reactive protein - hs-PCR levels evaluate the effect of periodontal therapy alone or with azithromycin on levels of high sensitivity C-reactive protein (hs CRP) in patients with chronic periodontitis

SECONDARY OUTCOMES:
STUDY ON THE EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER LIPIDIC PROFILE | 3 months
  evaluate the effect of periodontal therapy alone or with azithromycin on levels of profile lipidic (Total cholesterol, triglycerides, HDL, LDL) in patients with chronic periodontitis
STUDY ON THE EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER GLYCEMIA LEVELS | 3 months
  evaluate the effect of periodontal therapy alone or with azithromycin on levels of glycemia in patients with chronic periodontitis
STUDY ON THE EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER BLOOD BIOCHEMISTRY | 3 MONTHS
  evaluate the effect of periodontal therapy alone or with azithromycin on blood biochemistry (arterial index, hemogram) in patients with chronic periodontitis.

OTHER OUTCOMES:
STUDY ON THE EFFECTS OF PERIODONTAL TREATMENT ALONG WITH THE USE OF ANTIBIOTICS OVER PERIODONTAL PARAMETERS | 3 months
  evaluate the effect of periodontal therapy alone or with azithromycin on periodontal parameters (probing deep, bleeding on probing, clinical atachment level) in patients with chronic periodontitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Del Valle, Cali, Colombia